CLINICAL TRIAL: NCT00718289
Title: Citrate- Versus Acetate-Based Dialysate in Bicarbonate Haemodialysis: Consequences on Haemodynamics, Coagulation, Acid-Base Status and Electrolytes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Regionale di Locarno (Other)
Collaborators: Bichsel AG, Interlaken, Switzerland (Unknown)
Responsible Party: Luca Gabutti; Head of Department, Ospedale Regionale di Locarno
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 012008
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Haemodialysis
Keywords: Citric acid; citrate; acetic acid; acetate; haemodialysis; calcium; hypotension; haemodynamics; Dialysate for Haemodialysis
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citrate (Experimental): Citrate dialysate for haemodialysis
  Interventions: Other: Citrate dialysate
- Acetate (Active Comparator): Acetate dialysate
  Interventions: Other: Acetate dialysate

INTERVENTIONS:
Other: Citrate dialysate — dialysis fluid composition for Citrate (C) and Acetate (A): acetate [3.0 mmol/L in A and 0.3 in C], citrate [0 mmol/L in A and 0.8 in C]
  Arms: Citrate
Other: Acetate dialysate — dialysis fluid composition for Citrate (C) and Acetate (A): acetate [3.0 mmol/L in A and 0.3 in C], citrate [0 mmol/L in A and 0.8 in C]
  Arms: Acetate

SUMMARY:
Background:

A concentrate for bicarbonate haemodialysis acidified with citrate instead of acetate has been marketed in the recent years. The small amount of citrate used (one-fifth of the concentration adopted in regional anticoagulation) protects against intradialyser clotting, minimally affecting the calcium concentration. The aim of this study is to compare the impact of a citrate- and acetate-based dialysate on systemic haemodynamics, coagulation, acid-base status, calcium balance and dialysis efficiency.

Methods:

In 25 patients, 375 dialysis sessions, we will compare acetate (A) with citrate dialysate with (C+) or without (C) calcium supplementation (0.25mmol/L) in a randomized single blind cross-over study. Systemic haemodynamics will be evaluated using pulse wave analysis systems. Coagulation, acid-base status, calcium balance and dialysis efficiency will be assessed using standard biochemical markers.

DETAILED DESCRIPTION:
Introduction:

A concentrate for bicarbonate haemodialysis acidified with citric instead of the less physiologic acetic acid has been successfully implemented in the United States in the past 7 years [1-3]. Contrarily to traditional regional citrate anticoagulation, the small amount of citrate used in the acid concentrate (0.8 mmol/L only; about one-fifth of the concentration necessary to achieve anticoagulation [1,4,5]) affects the calcium concentration and the locally enhanced coagulation activation in a limited way, resulting in approximately 10% reduction in post-dialysis ionized calcium and in no measurable systemic anticoagulation [1]. The absence of significant systemic repercussions is related to both, the low amount of citrate used but also the rapid conversion of citrate into bicarbonate taking place in the liver and muscles and determining a higher post-dialysis bicarbonataemia [1,6,7]. Despite the rapid citrate clearance, the local consequences of removing calcium from the blood clotting cascade has measurable positive effects on the dialyser life-span in the "reuse" modality and on the dialysis quality quantified by urea Kt/V [1,3]. The improvement in urea clearance was correlated to a postulated favourable effect on dialyser fibre permeability mediated by the intra-dialyser anticoagulants properties of citrate [1,3,8]. Considering the importance of limiting the biocompatibility related coagulation activation taking place in the extracorporeal circuit [9-17], disposing of a simple way to inhibit it without affecting the systemic coagulation and the bleeding risk [18] is very promising.

Even if thousands of patients have been treated in the recent years with haemodialysis fluids based on citric instead of acetic acid, the haemodynamic tolerance (the reduction in ionized calcium concentration and the increase in bicarbonateamia could both result in a lower intra-dialytic blood pressure [19-25]) and the amount of systemic coagulation activation related to each one of the modalities, were not investigated.

The aim of this randomized, controlled, single blind, cross-over study in single-use dialyser bicarbonate haemodialysis, is to detail the consequences on systemic haemodynamics, coagulation activation, acid-base status, calcium balance and dialysis efficiency of using citric instead of acetic acid in the haemodialysis fluids.

Methods and patients:

Twenty-five chronic haemodialysis patients (15 male and 10 female), dialysed 3 to 4 hours three times a week, clinically stable and without intercurrent illnesses, will be enrolled in the study. Using a single blind, cross-over design, the patients will be randomized in the two arms of the study beginning by either the traditional acetic acid (modality A) or the citric acid dialysate (modality C). In the following 3 weeks the modality will be weekly switched to the alternative one. Finally, with the intention to compensate the reduction in serum calcium induced by the citrate binding, both study arms will be completed with a week using a citric acid dialysate with a calcium supplementation of 0.25 mmol/L (modality C+).

The haemodialyses will be performed using a 4008 H machine, equipped with a cartridge of bicarbonate Bibag©, and a high flux single use polysulfone membrane, all from Fresenius Medical Care (Bad Homburg, Germany). The prescribed dialyser effective surface area, dialysis fluid conductibility, temperature and composition (with the exception of acetate [3.0 mmol/L in A and 0.3 in C and C+], citrate [0 mmol/L in A and 0.8 in C and C+] and calcium [1.25 and 1.50 mmol/L in A and C and 1.50 and 1.75 in C+]), and effective blood flow will be recorded at the enrolment in the study, and left unchanged for the following 5 weeks. The medications of the patients (including phosphate binders) will also be left unchanged.

Serum BUN, creatinine, potassium, phosphate, calcium and whole blood pH, bicarbonate, and ionized calcium will be measured at the beginning and at the end of the third dialysis session of each week. Ionized and total calcium will also be measured at the beginning and at the end of the first dialysis session of each week. The prothrombin fragments 1+2 (F1+2) and thrombin-antithrombin complexes (TAT) will be determined at the beginning and at the end of the third dialysis session of each week [26]. Blood samples will be taken from the arterial limb of the shunt.

Systolic and diastolic blood pressures and heart rate will be measured before starting every session, and then repeated at 30 min interval throughout the dialysis with an automated Blood Pressure Monitor 4008 (Fresenius Medical Care, Bad Homburg, Germany) integrated in the dialysis machine. Stroke volumes (integrated mean of the flow waveform between the current upstroke and the dicrotic notch) and peripheral resistances (ratio of mean arterial pressure to stroke volume multiplied by heart rate) will be evaluated between 5 and 10 minutes after starting the session and then every 45 minutes using a finger beat-to-beat monitor Finometer© (Finapres Medical Systems BV, Arnhem, The Netherlands). The use of isotonic saline (100-200 ml) infusions to treat symptomatic hypotension or symptoms related to intravascular hypovolaemia will be registered.

Kt/V will be calculated using a second generation single-pool Daugirdas formula (Kt/V = -ln(R-0.03) + [(4-3.5 x R) x (UF/W)] where R = post-dialysis BUN/pre-dialysis BUN, UF = net ultrafiltration and W = weight).

The citrate accumulation during dialysis will be estimated calculating the calcium gap = │post-predialysis total calcium│- │post-predialysis ionized calcium│[6]. The value of 0.2 mmol/L will be used as a cut-off to divide the patients in rapid (< 0.2 mmol/L) and slow (≥ 0.2 mmol/L) metabolizers.

Results will be expressed as mean ± SD. Statistical analyses will be performed using a statistical software package (SPSS 12.0; SPSS Inc., Chicago, IL, USA). Comparisons between laboratory and haemodynamic parameters will be done first with an ANOVA followed if significant by a paired t-test performed between the mean of the values obtained in each patient with each modality. Haemodynamic parameters as a function of the dialysis time will be compared using a trapezoidal estimation of the area under the curves followed by a Wilcoxon Signed Ranks test. With the intention of ameliorating the understanding of the haemodynamic changes, an evaluation of the maximum increase and decrease in each parameter will be added to the data analysis (see Figure 2 for an explanation of the calculation method). Percentages will be compared using a Fisher Exact test. In all cases, a P ≤ 0.05 will be considered statistically significant; P will be expressed as ns (not significant), =0.05, <0.05, <0.01 and <0.001.

The protocol of the study has been approved by the local Ethical Committee. All the patients will give written informed consent prior to enrolment in the study.

References:

1. Ahmad S, Callan R Cole JJ, Blagg CR. Dialysate made from dry chemicals using citric acid increases dialysis dose. Am J Kidney Dis. 2000;35,493-499.
2. Tu A, Ahmad S. (2000). Heparin-free hemodialysis with citrate-containing dialysate in intensive care patients. Neph Dial Transplant. 2000;29,620-626.
3. Ahmad S, Callan R, Cole J, Blagg C. Increased dialyzer reuse with citrate dialysate. Hemodial Int. 2005;9:264-267.
4. Apsner R, Buchmayer H,Gruber D, Sunder-Plassmann G. Citrate for long-term hemodialysis: prospective study of 1,009 consecutive high-flux treatments in 59 patients. Am J Kidney Dis. 2005;45:557-564.
5. Pinnick RV, Wiegmann TB, Diederich DA. Regional citrate anticoagulation for hemodialysis in the patient at high risk for bleeding. N Engl J Med. 1983;308:258-61.
6. Bauer E, Derfler K, Joukhdar C, Druml W. Citrate kinetics in patients long-term hemodialysis therapy.Am J Kidney Dis. 2005;46:903-907.
7. Gabutti L, Marone C, Colucci G, Duchini F, Schönholzer C. Citrate anticoagulation in continuous venovenous hemodiafiltration: a metabolic challenge. Intensive Care Med. 2002;28,1419-1425.
8. Gabutti L, Colucci G, Martella A, Schönholzer C, Marone C. Does monitoring of pre-/post-dialyzer pressure difference improve efficiency in intermittent hemodialysis ? Blood Purif. 2003;21,294-300.
9. Gabutti L, Ferrari N, Mombelli G, Keller F, Marone C. The favorable effect of regional citrate anticoagulation on interleukin-1beta release is dissociated from both coagulation and complement activation. J Nephrol. 2004;17,819-825.
10. Stiekema JC. Heparin and its biocompatibility. Clin Nephrol. 1986;26:S3-8.
11. Cheung AK, Faezi-Jenkin B, Leypoldt JK. Effect of thrombosis on complement activation and neutrophil degranulation during in vitro hemodialysis. J Am Soc Nephrol. 1994;5:110-115.
12. Böhler J, Schollmeyer P, Dressel B, Dobos G, Hörl W. Reduction of granulocyte activation during hemodialysis with regional citrate anticoagulation: dissociation of complement activation and neutropenia from neutrophil degranulation. J Am Soc Nephrol. 1996;7:234-241.
13. Hofbauer R, Moser D, Frass M, Oberbauer R, Kaye AD, Wagner O, Kapiotis S, Druml W. Effect of anticoagulation on blood membrane interactions during hemodialysis. Kidney Int. 1999;56:1578-1583.
14. Bos JC, Grooteman MP, Van Houte AJ, Schoorl M, Van Limbeek J, Nube MJ. Low polymorphonuclear cell degranulation during citrate anticoagulation: a comparison between citrate and heparin dialysis. Nephrol Dial Transplant. 1997;12:1387-1393.
15. Dhondt A, Vanholder R, Tielemans C, Glorieux G, Waterloos MA, De Smet R, Lameire N. Effect of regional citrate anticoagulation on leukopenia, complement activation and expression of leukocyte surface molecules during hemodialysis with unmodified cellulose membranes. Nephron. 2000;85:334-342.
16. Bartels PC, Schoorl M, Wiering JG, Nube MJ. Activation of coagulation during treatment with hemodialysis. Scand J Clin Lab Invest. 2000;60:283-290.
17. Wiegmann TB, McDougall ML, Diederich DA. Dialysis leukopenia, hypoxemia and anaphylatoxin formation: effect of membrane, bath and citrate anticoagulation. Am J Kidney Dis 1988;11:418-424.
18. Fischer KG. Essentials of anticoagulation in hemodialysis.Hemodial Int. 2007;11:178-189.
19. Kaye M, Vasilevsky M, Ketis M. The effect on blood pressure of an acute fall in ionized calcium during hemodialysis. A randomized study in two patients. Clin Nephrol. 1998;50:361-366.
20. Van der Sande FM, Cheriex EC, Van Kuijk WHM, Leunissen KML. Effect of dialysate calcium concentrations on intradialytic blood pressure course in cardiac-compromised patients. Am J Kidney Dis. 1998;32:125-131.
21. Leunissen KML, Van den Berg BW, van Hooff JP. Ionized calcium plays a pivotal role in controlling blood pressure during haemodialysis. Blood Purif. 1989;7:233-239.
22. Sherman RA, Bialy GB, Gazinski B, Bernholc AS, Eisinger RP. The effect of dialysate calcium levels on blood pressure during hemodialysis. Am J Kidney Dis. 1986;8:244-247.
23. Maynard JC, Cruz C, Kleerekoper M, Levin NW. Blood pressure response to changes in serum ionized calcium during hemodialysis. Ann Intern Med. 1986;104:358-361.
24. Gabutti L, Ross V, Duchini F, Mombelli G, Marone C. Does Bicarbonate transfer have relevant hemodynamic consequences in standard hemodialysis? Blood Purif. 2005;23:365-372.
25. Gabutti L, Ferrari N, Giudici G, Mombelli G, Marone C. Unexpected haemodynamic instability associated with standard bicarbonate haemodialysis. Nephrol Dial Transplant. 2003;18:2369-2376.
26. Nossel HL, Yudelman I, Canfield RE, Butler VP, Spanondis K, Wilner GD, Qureshi GD. Measurement of fibrinopeptide A in human blood. J Clin Invest. 1974;54:43-53.

ELIGIBILITY:
Inclusion Criteria:

* chronic haemodialysis patients
* dialysed 3 to 4 hours three times a week, who were
* clinically stable and without intercurrent illnesses

Exclusion Criteria:

* intercurrent illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Consequences on systemic haemodynamics | Study duration

SECONDARY OUTCOMES:
Consequences on coagulation, acid-base status, calcium balance and dialysis efficiency | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gabutti, MD, Principal Investigator — Ospedale Regionale di Locarno
Locations (1):
- Ospedale Regionale di Locarno, Locarno, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Gabutti L, Lucchini B, Marone C, Alberio L, Burnier M. Citrate- vs. acetate-based dialysate in bicarbonate haemodialysis: consequences on haemodynamics, coagulation, acid-base status, and electrolytes. BMC Nephrol. 2009 Mar 5;10:7. doi: 10.1186/1471-2369-10-7. PMID 19265544